CLINICAL TRIAL: NCT06906523
Title: Blood Flow Restriction in Older Adults. A Randomised Single-blind Clinical Trial
Brief Title: Blood Flow Restriction in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Old-Rest
Record Dates: First submitted 2025-03-11; First posted 2025-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Older Patients
Keywords: Blood flow restriction; Older adults; Muscle power; Muscle strength; Functionality; Physical fitness
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (Experimental): An exercise protocol will be applied to work on lower limb strength in extension, with the application of BFR, with two 30-minute sessions per week for four weeks. The exercise protocol, based on previous studies in older adults, will consist of three exercises: climbing on a step, knee extension from a seated position and sitting down and getting up from a chair.
  Interventions: Other: Blood flow restriction training
- No intervention (No Intervention): Patients included in the control group will not receive any intervention, maintaining their activities of daily living in the same way as before the study.

INTERVENTIONS:
Other: Blood flow restriction training — The intensity of the work will be set at around 40% of the maximum intensity that can be executed in a single repetition (1RM). To reach the established intensity, weights, weighted ankle supports and rubber bands of different resistances will be used. Three sets of 8-10 repetitions will be performed with breaks of 1-2 seconds between repetitions and 2-3 minutes between sets. The intensity of the work will be established by applying the rate of perceived exertion. A blood flow restriction device will be used (Akrafit, Valencia, Spain model).
  Arms: Blood flow restriction

SUMMARY:
Introduction. From the age of 80 onwards, more than 50% of people suffer from sarcopenia. The loss of muscle strength leads to a loss of muscle power, impairing functionality and preventing the correct performance of activities of daily living.

Objective. To analyse the efficacy of blood flow restriction in older adult patients by evaluating changes in the variables muscle power and strength, physical condition and functionality of the lower limbs.

Material and method. Randomised single-blind clinical study. Thirty-six older adults will be recruited and randomised to the experimental and control groups. The intervention will have a duration of 4 weeks, with 2 weekly sessions. The intervention will consist of an intervention by performing 3 quadriceps strength exercises, with a 40% restriction. The primary variable of the study will be muscle power (Sit To Stand 5 times) and the secondary variables will be muscle strength (dynamometry), physical condition (Timed Up and Go) and functionality and autonomy (Barthel index)

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65 to 80 years
* Independent for standing and walking with the help of assistive devices such as cane and walker
* Both genders
* Normotensive or hypertensive with controlled BP (systolic blood pressure <140 mmHg)
* Sign the informed consent form.

Exclusion Criteria:

* People dependent for the performance of activities of daily living.
* People with cognitive impairments that limit the performance of the intervention or assessments.
* Persons undergoing total hip or knee arthroplasty
* Persons receiving physiotherapy treatment at the time of the study
* History of deep vein thrombosis (DVT) or pulmonary embolism
* History of myocardial infarction or stroke

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline muscle power after treatment and at four weeks | Screening visit, within the first seven days after treatment and four weeks follow-up visit
  Muscle power will be assessed with the Sit To Stand 5 times. This tool consists of getting up and sitting down from a chair five times. This instrument has shown high reliability (CCI= 0.95). The unit of measurement is time in seconds, where the shorter the time the greater the muscle power

SECONDARY OUTCOMES:
Change from baseline muscle strength after treatment and at four weeks | Screening visit, within the first seven days after treatment and four weeks follow-up visit
  Muscle strength shall be measured with a pressure dynamometer (Lafayette Manual Muscle Tester 01165). For the measurement of quadriceps muscle strength, the patient shall be placed in a seated position with 90° hip flexion and 75° knee flexion. The dynamometer shall be placed perpendicular to the leg to be assessed, just above the lateral malleolus, maintaining 75° of knee flexion. This assessment has shown good intra-observer reliability (ICC>0.70). This device measures in Newton the force performed by the patient in the requested muscle action. The higher the value, the greater the muscle strength
Change from baseline physical condition after treatment and at four weeks | Screening visit, within the first seven days after treatment and four weeks follow-up visit
  Physical condition will be measured with the Timed Up and Go (TUG). This tool consists of the participant getting up from a chair, walking three metres around an obstacle, walking back to the chair and sitting down again in a timed manner. This instrument has shown high reliability (ICC=0.80-0.99). The unit of measurement is time in seconds, where the shorter the time the greater the physical condition
Change from baseline functionality after treatment and at four weeks | Screening visit, within the first seven days after treatment and four weeks follow-up visit
  Functionality and autonomy will be measured with the Barthel Index. This tool consists of a scale assessing ten items: eating, transferring between chair and bed, personal grooming, toilet use, bathing/showering, transferring, going up and down stairs, dressing and undressing, stool control and urine control. Each item is scored 0 (dependent), 5 (performs with assistance) or 10 (independent) according to the degree to which he/she is able to perform it. This instrument has shown high reliability (ICC= 0.96). The score range is from 0 (total dependence) to 100 (independence).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No